CLINICAL TRIAL: NCT02571504
Title: Brain Imaging to Understand HIV-associated Neurocognitive Disorder and Predict Response to Cognitive Training
Brief Title: Cognitive Training for the Remediation of Functional Brain Health in HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Posit Science Corporation (Industry)
Responsible Party: Principal Investigator, Lesley K. Fellows, Neurologist, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 14-367 BMD; CTNPT 026 (Other: CIHR Canadian HIV Trials Network)
Record Dates: First submitted 2015-08-25; First posted 2015-10-08 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: HIV - Human Immunodeficiency Virus; Cognitive Impairment
Keywords: HIV - Human Immunodeficiency Virus; Memory; Concentration
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate cognitive training group (Experimental): Plasticity-based Adaptive Cognitive Remediation (PACR) is an 8 week training to improve executive functions (e.g., working memory, flexibility, cognitive control) as well as attention. Participants in the immediate cognitive training group will receive the PACR intervention shortly after enrollment.
  Interventions: Behavioral: Plasticity-based Adaptive Cognitive Remediation (PACR)
- Waitlist control group (Experimental): Participants in the waitlist control group will receive a brochure with 8 simple tips for better brain health around the time of enrollment. They will begin the Plasticity-based Adaptive Cognitive Remediation (PACR) intervention within 8 weeks of the initial enrollment.
  Interventions: Behavioral: Plasticity-based Adaptive Cognitive Remediation (PACR)

INTERVENTIONS:
Behavioral: Plasticity-based Adaptive Cognitive Remediation (PACR) — Web-based cognitive training program focused on improving attention and executive function (designed by Posit Science)

SUMMARY:
Cognitive deficits in HIV reflect degraded brain network functioning that may be amenable to remediation through cognitive training. In this sub-study, we will make use of Plasticity-based Adaptive Cognitive Remediation (PACR), which applies well-understood techniques derived from brain plasticity and implicit/procedural/perceptual learning to improve the speed and accuracy of information processing, with exercises that are designed to drive generalized improvements. Simultaneously, these exercises heavily engage neuromodulatory systems to re-establish their normal control over learning and memory. As an individual restores these degraded abilities through intensive procedural learning, the encoding of naturalistic information significantly improves, and all resulting declarative memory and cognitive functions based on the quality of that incoming information necessarily improve as well, leading to improvement that generalizes beyond the trained tasks.

A subset of 80 HIV+ individuals will undergo eight weeks of PACR to determine its feasibility and appropriateness for people with mild cognitive difficulties related to HIV infection. The results of this study are expected to be pivotal in generating data to create an optimal training program aimed at stabilizing or improving brain function in HIV infected individuals experiencing cognitive decline.

DETAILED DESCRIPTION:
The typical patterns of cognitive deficits in HIV reflect degraded brain network functioning, likely due to a combination of brain health insults: some generic (aging), some HIV-specific (inflammation, diffuse demyelination and inherent vulnerability that varies across individuals). Consistent with this view, the cognitive domains most affected are those that rely on extended networks (e.g. attention and executive functions relying on fronto-parietal and fronto-striatal circuits), exquisite timing (psychomotor function), or both. These network-based cognitive functions are vulnerable, but they are also resilient: there is a high degree of learning-dependent plasticity in networks involving the frontal lobes. This argues that the cognitive deficits in HIV may be amenable to remediation through cognitive training, and suggests mechanisms by which this might occur. There are many forms of cognitive rehabilitation; approaches that take advantage of advances in our understanding of the mechanisms of neuroplasticity and the neural systems supporting human cognition are likely to be highest yield. In this study, we will make use of Plasticity-based Adaptive Cognitive Remediation (PACR), a powerful method for harnessing this plastic potential. Conceptually, PACR applies well-understood techniques derived from brain plasticity and implicit/procedural/perceptual learning to improve the speed and accuracy of information processing, with exercises that are designed to drive generalized improvements. Simultaneously, these exercises heavily engage neuromodulatory systems to re-establish their normal control over learning and memory. As an individual restores these degraded abilities through intensive procedural learning, the encoding of naturalistic information significantly improves, and all resulting declarative memory and cognitive functions based on the quality of that incoming information necessarily improve as well, leading to improvement that generalizes beyond the trained tasks. Multiple randomized controlled studies have now demonstrated that PACR improves cognitive and functional abilities in patient populations with cognitive dysfunction similar in type and magnitude to patients with cognitive deficits due to HIV.

PACR runs in a web browser on any Internet connected computer and is implemented in an engaging game-like format. The participant selects one of the cognitive exercises scheduled for the day, and performs that exercise for fifteen minutes. The exercise itself contains the core science stimuli and task built into a game-like experience. Participants perform tens to hundreds of trials over the course of the fifteen-minute session, with each trial providing auditory and visual feedback and rewards to indicate if the trial was performed correctly or incorrectly. After each trial, the difficulty of the next trial is updated to ensure that within a session, the participant gets ~85% of trials correct. Thus, training is individually tailored to maximize its effectiveness. Summary screens including game metrics (points, levels) and exercise metrics (usage, progress) are shown to the participant at the end of each session. The scheduling mechanism ensures that a patient progresses through the exercises in a defined order, generally moving from more simple (early sensory processing) exercises to more complex (multimodal, cognitive control) exercises over the course of the 8 weeks experience. At any point in time, the participant only has access to a subset (typically six) of these exercises, four of which are performed per day.

Each exercise has specific criteria for completion, and after those criteria are met the exercise is removed from the active set and the next exercise added. This mechanism ensures both ongoing novelty and engagement for the participant, and that the participant progresses smoothly through the complete set of exercises over the program use period.

Free access will be provided to the PACR program, and a tailored cognitive training program will be developed in both French and English, specifically targeting domains and mechanisms that are most affected in HIV. This will include selection of the most suitable training modules (12 are planned), and optimization of the Web-based presentation and feedback to ensure acceptability to this target group.

The treatment goal will be use of the assigned program in 30 minutes sessions, five sessions per week, for 8 weeks after randomization; program use will be any mix of at home (or community Internet resource) or in-clinic sessions.

The outcome will be responder status (defined as improvement of >0.5 logits) on the B-CAM. With the assumption that the outcome is drawn from a binomial distribution with an expected probability of response of 10% (n=3) with no intervention, 30 subjects in the immediate training group will allow detection of a positive response at P<0.05 if 7 or more persons respond. The observed responses in both groups will provide more accurate estimates to plan for a scale up of this work to a full trial. An exploratory analysis will evaluate response in only those who completed at least 60% of the training sessions, recognizing that power here will be reduced, but the information nonetheless important.

Participants from both groups will also be compared to all those eligible for randomization to this intervention in the platform as a whole. Generalized estimating equations (GEE) will be applied as a secondary, more general approach here that permits other time points to be modeled, and consideration of other outcomes. This accommodates either binary (responder status) or continuous (scores on cognitive tests) outcomes. This analysis uses a regression model, but clustering of outcomes within time is controlled. For binary outcomes, the effect of group (immediate or control) is expressed as an odds ratio; for continuous outcomes the parameter is an effect size equivalent to an adjusted paired-t-test. An interaction term tests whether the effect differed by group (i.e. was larger in the immediate training group as hypothesized).

Additional analyses will be used to explain changes in B-CAM score as a function of changes expected from the intervention. As the intervention cohort is small, we will use concordance parameters, rather than a regression model, to quantify the degree to which changes in hypothesized mechanisms by which the interventions operate are concordant (at the individual level) with changes in the outcomes (cognitive ability).

ELIGIBILITY:
Inclusion Criteria:

* age 35 years or older;
* HIV infection for at least 1 year;
* able to communicate in English or French;
* capable of providing informed consent;
* easy access to the internet;
* EEG and MRI compatible

Exclusion Criteria:

* presence of dementia;
* life expectancy < 3 y;
* other neurological disorder including active opportunistic CNS infection;
* psychotic disorder;
* current substance dependence or abuse; and
* Hepatitis C requiring interferon therapy during the study period

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Brief Cognitive Ability Measure (B-CAM) | 3-4 months
  Ruler-like measure of cognitive ability combining self-report and performance items

SECONDARY OUTCOMES:
Change in Brain Health Indicators | 3 months
  Questionnaire on changes in self-report brain health indicators
Perceived Deficits Questionnaire | 9 months
  Questionnaire on changes in self-report cognitive concerns

CONTACTS AND LOCATIONS:
Overall Officials: Lesley K Fellows, MD, DPhil, Principal Investigator — McGill University
Locations (1):
- Montreal Neurological Institute and Hospital (McGill University), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymized individual data may be requested from the investigators.

REFERENCES:
- [Background] Clifford DB, Ances BM. HIV-associated neurocognitive disorder. Lancet Infect Dis. 2013 Nov;13(11):976-86. doi: 10.1016/S1473-3099(13)70269-X. PMID 24156898
- [Background] Power C, Boisse L, Rourke S, Gill MJ. NeuroAIDS: an evolving epidemic. Can J Neurol Sci. 2009 May;36(3):285-95. doi: 10.1017/s0317167100007009. PMID 19534327
- [Background] Au A, Cheng C, Chan I, Leung P, Li P, Heaton RK. Subjective memory complaints, mood, and memory deficits among HIV/AIDS patients in Hong Kong. J Clin Exp Neuropsychol. 2008 Apr;30(3):338-48. doi: 10.1080/13803390701416189. Epub 2007 Jul 25. PMID 17852611
- [Background] Holt JL, Kraft-Terry SD, Chang L. Neuroimaging studies of the aging HIV-1-infected brain. J Neurovirol. 2012 Aug;18(4):291-302. doi: 10.1007/s13365-012-0114-1. Epub 2012 Jun 1. PMID 22653528
- [Background] Vinogradov S, Fisher M, de Villers-Sidani E. Cognitive training for impaired neural systems in neuropsychiatric illness. Neuropsychopharmacology. 2012 Jan;37(1):43-76. doi: 10.1038/npp.2011.251. Epub 2011 Nov 2. PMID 22048465
- [Background] Mahncke HW, Bronstone A, Merzenich MM. Brain plasticity and functional losses in the aged: scientific bases for a novel intervention. Prog Brain Res. 2006;157:81-109. doi: 10.1016/S0079-6123(06)57006-2. PMID 17046669
- [Background] Fisher M, Holland C, Merzenich MM, Vinogradov S. Using neuroplasticity-based auditory training to improve verbal memory in schizophrenia. Am J Psychiatry. 2009 Jul;166(7):805-11. doi: 10.1176/appi.ajp.2009.08050757. Epub 2009 May 15. PMID 19448187
- [Background] Mahncke HW, Connor BB, Appelman J, Ahsanuddin ON, Hardy JL, Wood RA, Joyce NM, Boniske T, Atkins SM, Merzenich MM. Memory enhancement in healthy older adults using a brain plasticity-based training program: a randomized, controlled study. Proc Natl Acad Sci U S A. 2006 Aug 15;103(33):12523-8. doi: 10.1073/pnas.0605194103. Epub 2006 Aug 3. PMID 16888038
- [Background] Zelinski EM, Spina LM, Yaffe K, Ruff R, Kennison RF, Mahncke HW, Smith GE. Improvement in memory with plasticity-based adaptive cognitive training: results of the 3-month follow-up. J Am Geriatr Soc. 2011 Feb;59(2):258-65. doi: 10.1111/j.1532-5415.2010.03277.x. PMID 21314646
- [Background] Ances BM, Ortega M, Vaida F, Heaps J, Paul R. Independent effects of HIV, aging, and HAART on brain volumetric measures. J Acquir Immune Defic Syndr. 2012 Apr 15;59(5):469-77. doi: 10.1097/QAI.0b013e318249db17. PMID 22269799
- [Background] Tate DF, Conley J, Paul RH, Coop K, Zhang S, Zhou W, Laidlaw DH, Taylor LE, Flanigan T, Navia B, Cohen R, Tashima K. Quantitative diffusion tensor imaging tractography metrics are associated with cognitive performance among HIV-infected patients. Brain Imaging Behav. 2010 Mar;4(1):68-79. doi: 10.1007/s11682-009-9086-z. Epub 2010 Jan 19. PMID 20503115
- [Background] Du H, Wu Y, Ochs R, Edelman RR, Epstein LG, McArthur J, Ragin AB. A comparative evaluation of quantitative neuroimaging measurements of brain status in HIV infection. Psychiatry Res. 2012 Jul 30;203(1):95-9. doi: 10.1016/j.pscychresns.2011.08.014. Epub 2012 Aug 12. PMID 22892348
- [Background] Eskildsen SF, Coupe P, Garcia-Lorenzo D, Fonov V, Pruessner JC, Collins DL; Alzheimer's Disease Neuroimaging Initiative. Prediction of Alzheimer's disease in subjects with mild cognitive impairment from the ADNI cohort using patterns of cortical thinning. Neuroimage. 2013 Jan 15;65:511-21. doi: 10.1016/j.neuroimage.2012.09.058. Epub 2012 Oct 2. PMID 23036450
- [Background] Coupe P, Manjon JV, Fonov V, Pruessner J, Robles M, Collins DL. Patch-based segmentation using expert priors: application to hippocampus and ventricle segmentation. Neuroimage. 2011 Jan 15;54(2):940-54. doi: 10.1016/j.neuroimage.2010.09.018. Epub 2010 Sep 17. PMID 20851199
- [Background] Coupe P, Eskildsen SF, Manjon JV, Fonov VS, Collins DL; Alzheimer's disease Neuroimaging Initiative. Simultaneous segmentation and grading of anatomical structures for patient's classification: application to Alzheimer's disease. Neuroimage. 2012 Feb 15;59(4):3736-47. doi: 10.1016/j.neuroimage.2011.10.080. Epub 2011 Nov 9. PMID 22094645
- [Background] Jahanshad N, Valcour VG, Nir TM, Kohannim O, Busovaca E, Nicolas K, Thompson PM. Disrupted brain networks in the aging HIV+ population. Brain Connect. 2012;2(6):335-44. doi: 10.1089/brain.2012.0105-Rev. PMID 23240599
- [Background] Subramaniam K, Luks TL, Fisher M, Simpson GV, Nagarajan S, Vinogradov S. Computerized cognitive training restores neural activity within the reality monitoring network in schizophrenia. Neuron. 2012 Feb 23;73(4):842-53. doi: 10.1016/j.neuron.2011.12.024. PMID 22365555
- [Background] Sampaio-Baptista C, Scholz J, Jenkinson M, Thomas AG, Filippini N, Smit G, Douaud G, Johansen-Berg H. Gray matter volume is associated with rate of subsequent skill learning after a long term training intervention. Neuroimage. 2014 Aug 1;96:158-66. doi: 10.1016/j.neuroimage.2014.03.056. Epub 2014 Mar 26. PMID 24680712
- [Background] Concha L, Beaulieu C, Collins DL, Gross DW. White-matter diffusion abnormalities in temporal-lobe epilepsy with and without mesial temporal sclerosis. J Neurol Neurosurg Psychiatry. 2009 Mar;80(3):312-9. doi: 10.1136/jnnp.2007.139287. Epub 2008 Oct 31. PMID 18977826
- [Background] Tomaiuolo F, Scapin M, Di Paola M, Le Nezet P, Fadda L, Musicco M, Caltagirone C, Collins DL. Gross anatomy of the corpus callosum in Alzheimer's disease: regions of degeneration and their neuropsychological correlates. Dement Geriatr Cogn Disord. 2007;23(2):96-103. doi: 10.1159/000097371. Epub 2006 Nov 24. PMID 17127820
- [Background] He Y, Dagher A, Chen Z, Charil A, Zijdenbos A, Worsley K, Evans A. Impaired small-world efficiency in structural cortical networks in multiple sclerosis associated with white matter lesion load. Brain. 2009 Dec;132(Pt 12):3366-79. doi: 10.1093/brain/awp089. PMID 19439423
- [Background] Gauthier CJ, Desjardins-Crepeau L, Madjar C, Bherer L, Hoge RD. Absolute quantification of resting oxygen metabolism and metabolic reactivity during functional activation using QUO2 MRI. Neuroimage. 2012 Nov 15;63(3):1353-63. doi: 10.1016/j.neuroimage.2012.07.065. Epub 2012 Aug 16. PMID 22986357
- [Background] Lee EC, Whitehead AL, Jacques RM, Julious SA. The statistical interpretation of pilot trials: should significance thresholds be reconsidered? BMC Med Res Methodol. 2014 Mar 20;14:41. doi: 10.1186/1471-2288-14-41. PMID 24650044
- [Background] Sutton S, Braren M, Zubin J, John ER. Evoked-potential correlates of stimulus uncertainty. Science. 1965 Nov 26;150(3700):1187-8. doi: 10.1126/science.150.3700.1187. PMID 5852977
- [Background] Lesevre N. [Concepts underlying the analysis of late evoked potentials applied to the study of information processing and its disturbances in psychopathology]. Neurophysiol Clin. 1988 Feb;18(1):1-20. doi: 10.1016/s0987-7053(88)80103-5. French. PMID 3290642
- [Background] O'Brien JL, Edwards JD, Maxfield ND, Peronto CL, Williams VA, Lister JJ. Cognitive training and selective attention in the aging brain: an electrophysiological study. Clin Neurophysiol. 2013 Nov;124(11):2198-208. doi: 10.1016/j.clinph.2013.05.012. Epub 2013 Jun 14. PMID 23770088
- [Background] Tong Y, Melara RD, Rao A. P2 enhancement from auditory discrimination training is associated with improved reaction times. Brain Res. 2009 Nov 10;1297:80-8. doi: 10.1016/j.brainres.2009.07.089. Epub 2009 Aug 6. PMID 19651109
- [Background] Spironelli C, Bergamaschi S, Mondini S, Villani D, Angrilli A. Functional plasticity in Alzheimer's disease: effect of cognitive training on language-related ERP components. Neuropsychologia. 2013 Jul;51(8):1638-48. doi: 10.1016/j.neuropsychologia.2013.05.007. Epub 2013 May 14. PMID 23685197
- [Background] Okada YC, Kaufman L, Williamson SJ. The hippocampal formation as a source of the slow endogenous potentials. Electroencephalogr Clin Neurophysiol. 1983 Apr;55(4):417-26. doi: 10.1016/0013-4694(83)90130-x. PMID 6187535
- [Background] Goodin DS, Squires KC, Starr A. Long latency event-related components of the auditory evoked potential in dementia. Brain. 1978 Dec;101(4):635-48. doi: 10.1093/brain/101.4.635. PMID 737523
- [Background] Polich J, Kok A. Cognitive and biological determinants of P300: an integrative review. Biol Psychol. 1995 Oct;41(2):103-46. doi: 10.1016/0301-0511(95)05130-9. PMID 8534788
- [Background] Gevins A, Smith ME. Neurophysiological measures of working memory and individual differences in cognitive ability and cognitive style. Cereb Cortex. 2000 Sep;10(9):829-39. doi: 10.1093/cercor/10.9.829. PMID 10982744
- [Background] Goodin DS, Aminoff MJ, Chernoff DN, Hollander H. Long latency event-related potentials in patients infected with human immunodeficiency virus. Ann Neurol. 1990 Apr;27(4):414-9. doi: 10.1002/ana.410270409. PMID 2353795
- [Background] Gil R, Breux JP, Neau JP, Becq-Giraudon B. [Cognitive evoked potentials and HIV infection]. Neurophysiol Clin. 1992 Nov;22(5):385-91. doi: 10.1016/s0987-7053(05)80096-6. French. PMID 1484519
- [Background] Schroeder MM, Handelsman L, Torres L, Dorfman D, Rinaldi P, Jacobson J, Wiener J, Ritter W. Early and late cognitive event-related potentials mark stages of HIV-1 infection in the drug-user risk group. Biol Psychiatry. 1994 Jan 1;35(1):54-69. doi: 10.1016/0006-3223(94)91168-1. PMID 8167205
- [Background] Bauer LO. Interactive effects of HIV/AIDS, body mass, and substance abuse on the frontal brain: a P300 study. Psychiatry Res. 2011 Jan 30;185(1-2):232-7. doi: 10.1016/j.psychres.2009.08.020. Epub 2010 May 23. PMID 20580839
- [Background] Tartar JL, Sheehan CM, Nash AJ, Starratt C, Puga A, Widmayer S. ERPs differ from neurometric tests in assessing HIV-associated cognitive deficit. Neuroreport. 2004 Jul 19;15(10):1675-8. doi: 10.1097/01.wnr.0000134992.74181.4b. PMID 15232305
- [Background] Chao LL, Lindgren JA, Flenniken DL, Weiner MW. ERP evidence of impaired central nervous system function in virally suppressed HIV patients on antiretroviral therapy. Clin Neurophysiol. 2004 Jul;115(7):1583-91. doi: 10.1016/j.clinph.2004.02.015. PMID 15203059
- [Background] Baldeweg T, Gruzelier JH, Catalan J, Pugh K, Lovett E, Riccio M, Stygall J, Irving G, Catt S, Hawkins D. Auditory and visual event-related potentials in a controlled investigation of HIV infection. Electroencephalogr Clin Neurophysiol. 1993 Sep-Oct;88(5):356-68. doi: 10.1016/0168-5597(93)90012-e. PMID 7691560
- [Background] Toth B, File B, Boha R, Kardos Z, Hidasi Z, Gaal ZA, Csibri E, Salacz P, Stam CJ, Molnar M. EEG network connectivity changes in mild cognitive impairment - Preliminary results. Int J Psychophysiol. 2014 Apr;92(1):1-7. doi: 10.1016/j.ijpsycho.2014.02.001. Epub 2014 Feb 6. PMID 24508504
- [Background] van der Molen MJ, Stam CJ, van der Molen MW. Resting-state EEG oscillatory dynamics in fragile X syndrome: abnormal functional connectivity and brain network organization. PLoS One. 2014 Feb 11;9(2):e88451. doi: 10.1371/journal.pone.0088451. eCollection 2014. PMID 24523898
- [Background] Babiloni C, Vecchio F, Lizio R, Ferri R, Rodriguez G, Marzano N, Frisoni GB, Rossini PM. Resting state cortical rhythms in mild cognitive impairment and Alzheimer's disease: electroencephalographic evidence. J Alzheimers Dis. 2011;26 Suppl 3:201-14. doi: 10.3233/JAD-2011-0051. PMID 21971461
- [Derived] Mayo NE, Brouillette MJ, Fellows LK; Positive Brain Health Now Investigators. Understanding and optimizing brain health in HIV now: protocol for a longitudinal cohort study with multiple randomized controlled trials. BMC Neurol. 2016 Jan 14;16:8. doi: 10.1186/s12883-016-0527-1. PMID 26762403